CLINICAL TRIAL: NCT04803227
Title: Safety and Tolerability of Emricasan in Symptomatic Outpatients Diagnosed With Mild-COVID-19
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Unforeseeable difficulties in recruiting patients. There were no reported serious adverse events.
Sponsor: Histogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EMR-COV-PR001; www.pacestudies.com (Other: Histogen)
Record Dates: First submitted 2021-02-12; First posted 2021-03-17 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Covid19
Keywords: mild, symptomatic, COVID19
MeSH Terms: conditions — COVID-19; Lymphoma, Follicular | interventions — 3-(2-(2-tert-butylphenylaminooxalyl)aminopropionylamino)-4-oxo-5-(2,3,5,6-tetrafluorophenoxy)pentanoic acid

STUDY DESIGN:
Intervention Model Description: Double-blind, Placebo-controlled, Randomized, 1:1 active: placebo.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Emricasan (Active Comparator): Emricasan
  Interventions: Drug: Emricasan
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Emricasan — Emricasan 25 mg BID (days 1-14). Oral (capsule) administration.
  Arms: Emricasan
Other: Placebo — Placebo BID *days 1-14). Oral (capsule) administration.
  Arms: Placebo

SUMMARY:
Treatments for COVID-19 are urgently needed. Emricasan (EMR) is a pan caspase inhibitor. Caspase-1 plays a role in a form of cell death called pyroptosis. EMR inhibits pyroptosis. The Investigators have shown that peripheral blood lymphocytes of COVID-19 patients overexpress caspase-1, providing evidence for pyroptosis. A recent European study corroborate the Investigators finding as they have shown evidence for the activation of the inflammasome in COVID-19.

DETAILED DESCRIPTION:
A safety and tolerability study will be performed in 50 symptomatic outpatient mild-COVID-19 patients using Emricasan at 25mg BID dosing for 14 days with a 1:1 active: placebo of mild-COVID-19 patients receiving standard of care therapy. Although EMR has been extensively studied in humans in a total of 18 Phase 1 and Phase 2 studies, with an excellent safety and tolerance profile, it has not been used in the setting of COVID-19, therefore necessitating an initial safety and tolerability study looking at a no difference between AEs/SAEs for comparison between active and placebo group. The pharmacokinetics of EMR has been extensively studied; therefore, the Investigators will opportunistically sample patients at the end of the study to confirm that the Emricasan PK is not altered in COVID-19 patients. The primary endpoint will be cumulative incidence of AE/SAEs through day 14. Secondary endpoints will include various clinical and laboratory measures and patient reported outcomes (PROs) using a COVID-19-related assessment tool, SARS-CoV-2 viral PCR, titers of anti-SARS-CoV-2 neutralizing and quantitative antibodies and immunological studies as described in the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent form signed and dated by participant.
2. Men or women >/=18 years of age at the time of signing the informed consent.
3. Access to device and internet for Televisits.
4. Laboratory confirmed SARS-CoV-2 infection via viral RT-PCR test. The SARS-CoV-2 diagnostic test will be conducted using, if possible, an FDA acceptable product under Emergency use Authorization (EUA) or as cleared by the Center for Device and Radiological Health (CDRH). We will have confirmation of the SARS-CoV-2 testing prior to enrollment.
5. COVID-19 patients in generally healthy status without significant medical comorbidities.
6. A treatment window for first dose of up to 10 days from onset of symptoms.
7. Outpatients with symptoms of respiratory illness caused by coronavirus 2019 infection as defined below:

   * Symptoms of mild illness with COVID-19 as defined by the W.H.O. in Table 1of the Clinical Management of COVID-19 interim Guidance document, May 27, 2020, meeting the case definition for mild COVID-19 without evidence of viral pneumonia or hypoxia
   * COVID-19 severity score on an 8-point ordinal score =/< 2 as defined by the WHO

2020. 8. Clinically normal resting 12-lead ECG at Screening Visit or, if abnormal, considered not clinically significant by the Principal Investigator. 9. Normal or clinically insignificant change in the liver (ALT, AST) and kidney function (blood creatinine), CBC with differential and clotting factors (PT and PTT).

10. Understands and agrees to comply with planned study procedures. 11. Women of childbearing potential must agree to use at least one medically accepted method of contraception (e.g., barrier contraceptives [condom, or diaphragm with a spermicidal gel], hormonal contraceptives [implants, injectables, combination oral contraceptives, transdermal patches, or contraceptive rings], or intrauterine devices) for the duration of the study.

12. Background standard of care will be maintained in all treatment arms. Off-label use of any other drugs, devices, or interventions that might be used to manage COVID-19 need to be discussed with the study medical director.

Exclusion Criteria:

1. Subjects showing signs of acute respiratory distress syndrome (ARDS) or respiratory failure necessitating mechanical ventilation at the time of screening and ICU patients.
2. Patients with established COVID-19 co-morbidities, other than controlled hypertension, as established by current CDC-guidelines.
3. Unable to take oral medications.
4. Hospitalized patients at screening.
5. Moderate and severe hepatic impairment (Child-Pugh B and C) for phase 1 protocol.
6. History of severe chronic respiratory disease and requirement for oxygen therapy
7. Any uncontrolled active systemic infection (e.g. cellulitis or abscess) or infections requiring admission to an intensive care unit (ICU). Note: Subjects infected with HIV-1 will be eligible for the study with undetectable viral load and are on a stable ART regimen. Investigators are required to review the subjects' medical records to confirm HIV-1 RNA suppression within the previous 3 months.

   Note: Empirical antibiotic treatment for secondary bacterial infections is allowed during the course of study.
8. Patients with elevated baseline LFT's, such as an ALT / AST > 2 X ULN determined by the hospital lab.
9. Patients with diagnosed liver cirrhosis or clinical evidence suggestive of advanced liver disease.
10. Patients with malignant tumor(s), or other serious systemic diseases.
11. Patients who are participating in any other clinical studies.
12. Patients who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to leronlimab (PRO 140) are not eligible.
13. Current use of the following medications that are considered significant inhibitors of OATP1B1 and OATP1B3 transporters: atazanavir, cyclosporine, eltrombopag, gemfibrozil, indinavir, lopinavir, ritonavir, rifampin, saquinavir, simeprevir, telaprevir, tipranovir, or some combination of these medications
14. History or presence of clinically concerning cardiac arrhythmias, or prolongation of Screening (pre-treatment) QTcF interval >480 milliseconds (msec)
15. Inability to provide informed consent or to comply with test requirements
16. Moderate or higher level of severity of COVID-19. Moderate COVID-19 defined as: Symptoms of moderate illness with COVID-19, which could include any symptom of mild illness or shortness of breath with exertion, but clinical signs suggestive of moderate illness with COVID-19 including, respiratory rate ≥ 25 breaths per minute, or saturation of oxygen (SpO2) < 93% on room air at sea level, or resting heart rate ≥ 90 beats per minute (unless related to fever). In elderly patient population normal resting respiratory rate is 16-25 [24].
17. Immunocompromised patients and/or patients on immunomodulators or immune suppressants other than systemic or inhaled steroids, including transplant recipients.
18. Evidence of any new or uncontrolled concomitant disease that, in the investigator's judgment, would preclude patient participation, including but not limited to cardiovascular, pulmonary, nervous system, renal, hepatic, endocrine, malignant, or gastrointestinal disorders
19. If female, planned or known pregnancy - positive urine or serum pregnancy test
20. Lactating or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-05-28 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 14 Days
  Incidence rate of related treatment-emergent adverse events

SECONDARY OUTCOMES:
Patient reported outcomes as assessed by COVID-19 assessment tool | At screening/randomization, daily televisits (Day 2 - Day 13), Day 14, Day 30 and Day 45
  The 2020 FDA Guidance for Industry Assessing COVID-19-Related Symptoms in Outpatient Adult and Adolescent Subjects in Clinical Trials of Drugs and Biological Products for COVID-19 Prevention or Treatment is the PRO that will be used for the study.
Number of participants that experience death during the study. | 45 Days
  Rate of mortality events
Number of participants the experience a related serious adverse event as assessed by CTCAE v5.0. | 45 Days
  Cumulative incidence rate of related serious adverse events
Number of participants that experiences a Grade 3 and 4 adverse event as assessed by CTCAE v5.0 | 45 Days
  Cumulative incidence rate of Grade 3 and 4 adverse events
Number of participants with a discontinuation or temporary suspension of study drug | 45 days
  Each participant that discontinues or temporarily suspends study drug for any reason.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Day 1, Day 14, Day 30 and Day 45
  Each participant will be assessed via performance of standard of care hematology and biochemistry labs. The results of the labs will be assessed against a set of normal ranges for the CLIA certified laboratory.
Each participant will be tested for SARS-CoV-2 viral eradication via a sample from the nasopharynx and the sample will be tested via RT- PCR. | Days 14, 30 and 45
  SARS-CoV-2 viral eradication from nasopharynx at end of treatment.
Each participant will perform a 6 minute walk test (6MWD) for distance (400-700m) walked. | Days 14, 30 and 45
  Perform 6 Minute Walk Test
Each participant will be assessed for COVID-19 severity via an 8-point ordinal scale | Days 14, 30 and 45
  COVID-19 severity score on the 8-point COVID-19 Severity Scale. Scores are from 1 to 8, where 1 = uninfected and 8 = death
Each participant will be tested for anti-SARS-CoV-2 neutralizing antibodies via standard histogram, 2D plots, tSNE, and viSNE analysis. | Days 14, 30 and 45
  The following cell populations will be examined- NK, CD4 and CD8 T-cells, Tfh, Treg, CD4 and CD8 memory, B-cell memory, monocytes and dendritic cells.
Each participant will be tested for anti-SARS-CoV-2 quantitative antibodies via cytokine test panel. | Days 14, 30 and 45
  Immune test for titers of serum anti-SARS-CoV-2 quantitative antibodies
Each participant will be assessed for resolution of COVID19 symptoms via performance of hematology and biochemistry labs, SARS-COV-2 nasopharyngeal swab and tested via RT-PCR and immunology testing for cytokines and cell populations. | Days 14, 30 and 45
  Percentage of Participants with Resolution of COVID19 symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Raavi Gupta, MD, Principal Investigator — SUNY Downstate
Locations (1):
- SUNY Downstate Health Sciences University, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No